CLINICAL TRIAL: NCT05298085
Title: Effect of Intranasal Oxytocin on Dysphagia Related to Oropharyngo-oesophageal Dysmotility in Children and Adolescents With Prader-Willi Syndrome: a Phase 2B Study
Brief Title: Effect of Intranasal Oxytocin on Dysphagia in Children and Adolescents With Prader-Willi Syndrome
Acronym: DYSMOT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RC31/20/0518
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi syndrome; Oxytocin
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OXYTOCIN nasal spray (Experimental): intranasal administration of Oxytocin
  Interventions: Drug: Oxytocin nasal spray
- PLACEBO (Placebo Comparator): intranasal administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — Study treatment will be administered intranasally daily for 12 weeks. The daily dose of OT will be adapted according to age at the beginning of the study
  Other Names: oxytocin
  Arms: OXYTOCIN nasal spray
Drug: Placebo — Study treatment will be administered intranasally daily for 12 weeks.
  Other Names: placebo nasal spray
  Arms: PLACEBO

SUMMARY:
This phase 2B is designed to test the effectiveness of intranasal Oxytocin on Prader Willi Syndrome (PWS).

This is a prospective, multicentre, randomised, double-blind, Phase 2B clinical study planned to include around 24 PWS patients aged 2-17 years and 5 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 2 years and 17 years and 5 months at inclusion.
2. Genetically confirmed diagnosis of PWS.
3. Parents (or legal representative) have signed the informed consent form and are willing to comply with all study procedures.

Exclusion Criteria:

1. A history of hypersensitivity to the study drug or drugs with similar chemical structures, to excipients of the product, or to latex;
2. Intolerance of intranasal administrations (including when due to a major behavioural problem);
3. Hyponatremia (clinically relevant at the discretion of the investigator);
4. Hypokalaemia (clinically relevant at the discretion of the investigator);
5. Prolongation of the QT interval and/or family history of prolongation of the QT interval;
6. Concomitant treatment prolonging the QT interval;
7. Start of growth hormone (GH) treatment within the last 4 weeks before inclusion;
8. History of abnormal electrocardiogram (ECG) (validated by a cardiologist);
9. Pregnant girls; (for girls with childbearing potential who do not have contraception and are sexually active, a negative pregnancy test will be required)
10. Patient with clinical signs in the context of contact with COVID-19 infected person.
11. Patient included in another study protocol on a medicinal product within the last 6 months;
12. Administrative problems:

    1. Inability to give parents (or legal representatives) expert medical information;
    2. No coverage by a social security regime.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
videofluoroscopic swallowing study (VFSS) score change | after 12 weeks oxytocin (OT) / placebo (at V2)
  Percentage of patient with at least one VFSS subscore's change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: TAUBER Maithé, MD, Principal Investigator — University Hospital, Toulouse
Locations (4):
- France (4):
  - Hopital Jeanne de Flandre, Lille
  - Hôpital Femme-Mère-enfant Groupement hospitalier Est, Lyon
  - Chu Rouen, Rouen
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No